CLINICAL TRIAL: NCT01187576
Title: A Multi-professional Team Intervention on Physical Activity Referrals in Primary Care Patients With Cardiovascular Risk factors-the Dalby Lifestyle Intervention Cohort Study (DALICO) Study
Brief Title: A Multi-professional Team Intervention on Physical Activity Referrals in Primary Care Patients With Cardiovascular Risk Factors-the Dalby Lifestyle Intervention Cohort (DALICO) Study
Acronym: DALICO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started
Sponsor: Region Skane (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPF FaR 001
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Motivation for Physical Activity
Keywords: Physical activity; Hypertension; Diabetes mellitus; Motivational interviewing
MeSH Terms: conditions — Motor Activity; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention (Experimental): Multi-professional team intervention with PAR, lifestyle brochure
  Interventions: Behavioral: Multi-professional team intervention with PAR, lifestyle brochure
- Conventional treatment (Active Comparator): Ordinary recommendations on health behaviours, lifestyle brochure
  Interventions: Behavioral: Ordinary recommendations on health behaviours, lifestyle brochure
- retrospective med history comparison (No Intervention): Treatment as usual (retrospective data collection)

INTERVENTIONS:
Behavioral: Multi-professional team intervention with PAR, lifestyle brochure — Multi-professional team intervention with PAR, lifestyle brochure
  Arms: Intervention
Behavioral: Ordinary recommendations on health behaviours, lifestyle brochure — Ordinary recommendations on health behaviours, lifestyle brochure
  Arms: Conventional treatment

SUMMARY:
Background The present study protocol describes the trial design of a primary care intervention cohort study, which examines whether an extended, multi-professional physical activity referral (PAR) intervention is more effective in enhancing and maintaining self-reported physical activity than ordinary physical activity recommendations. The study targets patients with newly diagnosed hypertension and/or type 2 diabetes.

Secondary outcomes include: need of pharmacological therapy; blood pressure/plasma glucose; physical fitness and anthropometric variables; mental health; health related quality of life; and cost-effectiveness. Methods/Design The study is designed as a long-term intervention. Three primary care centres are involved in the study, each constituting one of three treatment groups: 1) Intervention group (IG): multi-professional team intervention with PAR, lifestyle brochure; 2) Control group A (CA): ordinary recommendations on health behaviours, lifestyle brochure; and 3) Control group B: treatment as usual (retrospective data collection).

The intervention is based on self-determination theory and follows the principles of motivational interviewing. Physical activity is measured with the International Physical Activity Questionnaire (IPAQ) and expressed as metabolic equivalent of task (MET)-minutes per week. Physical fitness is estimated with the 6-minute walk test in IG only. Variables such as health behaviours; health-related quality of life; motivation to change; mental health; demographics and socioeconomic characteristics are assessed with an electronic study questionnaire that submits all data to a patient database, which automatically provides instant feed-back on the patients' health status.

Cost-effectiveness of the intervention is evaluated continuously and the intermediate

- 3 - outcomes of the intervention are extrapolated by economic modelling. The first statistical analyses and compilation of results will be performed one year after inclusion of the first patient or when the IG and CA have included 60 and 30 eligible patients respectively. Discussion By helping patients to overcome practical, social and cultural obstacles and increase their internal motivation for physical activity we aim to improve their physical health in a long-term perspective. The targeted patients belong to a patient category that is supposed to benefit from increased physical activity in terms of improved physiological values, mental status and quality of life, decreased risk of complications and maybe a decreased need of medication.

ELIGIBILITY:
Inclusion Criteria:newly diagnosed type 2 diabetes or hypertension or both and consecutive primary care patients with suspected type 2 diabetes or hypertension will be screened for inclusion. The diagnose criterion for type 2 diabetes in both the Intervention and the Control groups is defined as a 2 x fasting plasma glucose (fP-glu) ≥ 7.0 mmol/l according to WHO guidelines [29]. The diagnose criterion for hypertension is defined as a resting systolic blood pressure ≥ 140 mmHg or a diastolic blood pressure ≥ 90 mmHg. Hypertension is confirmed by a 24-hour ambulatory blood pressure monitoring: a systolic blood pressure ≥ 135 mmHg and/or a

* 13 - diastolic blood pressure ≥ 85 mmHg

Exclusion Criteria:

-

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
to examine whether an extended multi-professional PAR intervention, based on SDT, is effective in increasing and maintaining the self-reported physical activity level in patients with newly diagnosed type 2 diabetes or hypertension or both. | every 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dalby Vårdcentral, Dalby, Sweden